CLINICAL TRIAL: NCT06028698
Title: Effects of Music on Table Tennis Stroke Performance Among Mentally Fatigued University Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ding Cong (Other)
Responsible Party: Sponsor-Investigator, Ding Cong, Principal Investigator, Universiti Putra Malaysia
Organization: Universiti Putra Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DingCong
Record Dates: First submitted 2023-08-24; First posted 2023-09-08 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Mental Fatigue
MeSH Terms: conditions — Mental Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Positive emotion music fatigue group (Experimental): After mental fatigue inducement, participants will be instructed listening to music pieces for inducing positive emotion music.
  Interventions: Other: Inducing positive emotion music
- Fatigue control group (Placebo Comparator): After mental fatigue inducement, participants will be instructed to sit and relax for the same duration as intervention group.
  Interventions: Other: Inducing positive emotion music
- No Fatigue positive emotion music group (Placebo Comparator): participants will not be induced mental fatigue, but will be instructed listening to music pieces for inducing positive emotion music.
  Interventions: Other: Inducing positive emotion music
- No fatigue control group (No Intervention): participants will not be induced mental fatigue. Also, participants will not receive music intervention，just sit and relax.

INTERVENTIONS:
Other: Inducing positive emotion music — listening to music could induce emotion response, this study is going to investigate inducing positive emotion music countering mental fatigue.
  Arms: Fatigue control group; No Fatigue positive emotion music group; Positive emotion music fatigue group

SUMMARY:
The current study is going to investigate the music intervention on the table tennis stroke performance among table tennis stroke performance. The subjects will be instructed to listen to 3 minutes, which can facilitate the recovering process for scope of attention and thought-action repertoire. Thus, to see the improvement in stroke performance.

DETAILED DESCRIPTION:
The intervention of this study is music, specifically, instruct subjects to listen inducing positive emotion music due to positive emotion benefit to cognition performance.

The condition of mental fatigue will be induced by Stroop task. Before the intervention or process of listening music, the pre-test will be recorded to compare the post-test value of table tennis stroke performance.

Moreover, the different music intervention will be implemented to identify the optimal selection.

ELIGIBILITY:
Inclusion Criteria:

* University table tennis players. 18-24 years.
* Both pen-holder and shake-hand play styles.
* At least played from the senior school.
* At least have 3 years' training experience.

Exclusion Criteria:

* Color blindness.
* Any disease or sleep disorder.
* Smoker or drunker

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
table tennis stroke performance | 4 weeks
  Before and after the intervention, stroke performance will be measured to see the difference. the stroke performance will be calculate based on formula: PI=Average speed × ball accuracy， the higher scores，the better stroke performance will be.
Ball speed | 4 weeks
  Before and after the intervention, ball speed will be measured to see the differences. the instrument of ball speed will be High speed camera, then input the videos into software Kinovea for measuring the fast speed
Ball accuracy | 4 weeks
  Before and after the intervention, ball accuracy will be measured to see the differences. the instrument of ball speed will be target position, for scoring 0-2 scores.

SECONDARY OUTCOMES:
Emotion state | 4 weeks
  Emotional state will be measured by Emotion Report Forms subjectively. This form consists of nine items, which are: Amusement, Anger, Anxiety, Contentment, Disgust, Fear, Happiness, Sadness, and Serenity, rated on a 9-point Likert scale. Participants report that higher scores represent a stronger current emotional state. A higher score for positive emotion items indicate a higher level of positive emotion was induced. The emotional state will be measured in baseline(before inducing mental fatigue); before and after the music intervention to observe any differences.
Scope of attention | 4 weeks
  Scope of attention will be measured by Global-local Processing Task, total 8 sets of stimulation. In each stimulation, participants will be instructed to select one figure (base on global configuration aspect or the local elements),which is more similar compare the the Standard figure. The more selection based on the global configuration by participants, means the more breadth of attention. Scope of attention will be measured in baseline(before inducing mental fatigue); before and after the music intervention to observe any differences.
Thought-action repertoire | 4 weeks
  Thought-action repertoire will be measured by Twenty Statement Test. Participants will be encouraged to fill the twenty blanks with:"i would like to " as many as possible, the more blanks filled by participants, the more score will be reported. the higher scores mean the more breadth of thought-action repertoire. Thought-action repertoire will be measured in baseline(before inducing mental fatigue); before and after the music intervention to observe any differences.

CONTACTS AND LOCATIONS:
Locations (1):
- Cong Ding, Huai'an, Jiangsu, China